CLINICAL TRIAL: NCT02508376
Title: A Phase 1, Randomized, Double Blind Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of the Vaccine Candidates ID93 + AP10-602 and ID93 + GLA-SE Administered Intramuscularly in Healthy Adult Subjects
Brief Title: Safety, Tolerability, and Immunogenicity of the Vaccine Candidates ID93 + AP10-602 and ID93 + GLA-SE Administered Intramuscularly in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12-0109; HHSN272201300020I
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-04-05

CONDITIONS: Tuberculosis
Keywords: adjuvants; AP10-602; GLA-SE; ID93; Tuberculosis; vaccine
MeSH Terms: conditions — Tuberculosis | interventions — glucopyranosyl lipid-A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ID93 (10 mcg) + AP10-602 (10 mcg) (Experimental): N=20 subjects will receive intervention on Days 1, 29, 57
  Interventions: Other: AP10-602; Biological: ID93
- ID93 (10 mcg) + AP10-602 (5 mcg) (Experimental): N=20 subjects will receive intervention on Days 1, 29, 57
  Interventions: Other: AP10-602; Biological: ID93
- ID93 (10 mcg) + GLA-SE (5 mcg) (Experimental): N=20 subjects will receive intervention on Days 1, 29, 57
  Interventions: Biological: GLA-SE; Biological: ID93
- ID93 (10 mcg) alone (Experimental): N=10 subjects will receive intervention on Days 1, 29, 57
  Interventions: Biological: ID93

INTERVENTIONS:
Other: AP10-602 — AP10-602 contains GLA formulated with liposomes and an additional immunological adjuvant. The ID93 (10 mcg) + AP10-602 (5 mcg) arm will receive intervention on days 1, 29 and 57. The ID93 (10 mcg) + AP10-602 (10 mcg) arm will receive intervention on days 1, 29 and 57.
  Arms: ID93 (10 mcg) + AP10-602 (10 mcg); ID93 (10 mcg) + AP10-602 (5 mcg)
Biological: GLA-SE — Glucopyranosyl Lipid A- Stable oil-in-water emulsion (GLA-SE). The ID93 (10 mcg) + GLA-SE (5 mcg) arm will receive intervention on days 1, 29 and 57
  Arms: ID93 (10 mcg) + GLA-SE (5 mcg)
Biological: ID93 — ID93 is a fusion polyprotein comprising four Mtb antigens (Rv2608, Rv3619, Rv3620, Rv1813). All arms will receive 10 mcg ID93 IM on days 1, 29 and 57

SUMMARY:
This is a phase I randomized, double blind clinical trial designed to evaluate the safety, tolerability and immunogenicity of the ID93 recombinant protein antigen alone or formulated with GLA-SE or AP10-602 adjuvant in 70 healthy adults 18-49 years of age. Subjects will receive a total of 3 doses administered intramuscularly on Days 1, 29 and 57. Subjects will be monitored for approximately 422 days (365 days following the third study injection), including safety laboratory analyses done just prior to and 7 days following each study injection. Blood samples will be obtained for immunological assays (Luminex, intracellular cytokine staining at Days 1 and 71, and antibody analysis at Days 1 and 85). The primary objective is to evaluate the safety and tolerability of 10 µg ID93 + 5 or 10 µg AP10-602 compared to 10 µg ID93 + 5 µg GLA-SE and 10 µg ID93 alone following three consecutive intramuscular injections administered on Days 1, 29 and 57.

DETAILED DESCRIPTION:
TB causes significant morbidity and mortality throughout the world. Strains of Mtb are becoming increasingly resistant to antimycobacterial drugs and therapy is often associated with poor compliance, which increases the likelihood of antimicrobial resistance. The current licensed BCG vaccine does not prevent reactivation or reinfection in adults so there is a great need for a more effective vaccine. ID93 is a recombinant antigen that, when mixed with the adjuvants GLA-SE and AP10-602, shows great promise in eliciting what is thought to be an important Th1 T cell response and limits the bacterial burden in Mtb challenged animals. This study is a phase I randomized, double blind clinical trial designed to evaluate the safety, tolerability and immunogenicity of the ID93 recombinant protein antigen alone or formulated with GLA-SE or AP10-602. This study will enroll 70 healthy males and non-pregnant females subjects, aged 18 to 49. Subjects who meet all eligibility criteria will be randomized to ID93 alone, ID93 + GLA-SE, or ID93 + AP10-602 at either dose level. Study injections will be performed and subjects will be observed in clinic for 30 minutes. All subjects will complete a written subject memory aid that solicits local and systemic reactogenicity adverse events for 7 days following each study injection. After subjects are reevaluated to ensure they continue to meet eligibility criteria they will undergo second and third study injections on Days 29 and 57. General safety will be evaluated on Days 1, 3, 8, 29, 31, 36, 57, 59, 64, 71, 85, 169, and 422 for each subject. The occurrence of serious adverse events and the new onset of any adverse events of special interest (AESI) will be collected throughout the study period (approximately 422 days). Each subject's duration of participation will be about 15 months. The Primary Objective is : To evaluate the safety and tolerability of 10 µg ID93 + 5 or 10 µg AP10-602 compared to 10 µg ID93 + 5 µg GLA-SE and 10 µg ID93 alone following three consecutive intramuscular injections administered on Days 1, 29 and 57. The Secondary Objective is: To assess the immunogenicity of 10 µg ID93 + 5 or 10 µg AP10-602 compared to 10 µg ID93 + 5 µg GLA-SE and 10 µg ID93 alone by quantifying T cell responses and IgG antibody responses to ID93 at specified time points.

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females between the ages of 18 and 49 years, inclusive. 2. Women of childbearing potential* must agree to practice adequate contraception** for the 28-day period before Day 0 through 90 days after the third study injection. * A woman is considered of childbearing potential unless surgically sterile (tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal (>/=1 year). **Acceptable birth control methods include but are not limited to: abstinence from sexual intercourse with men; monogamous relationship with a vasectomized partner; barrier methods (condoms, diaphragms, spermicides, and intrauterine devices); and licensed hormonal methods. 3. In good health, as judged by the investigator and determined by vital signs*, medical history, and a targeted physical examination. * Temperature <38°C, heart rate </=100 bpm and >54 bpm, systolic blood pressure </=140 mmHg and >89 mmHg, diastolic blood pressure </=90 mmHg and >/=60 mmHg. NOTE: Athletically trained subjects with a pulse >/=45 may be enrolled at the discretion of the principal investigator or designated licensed clinical investigator. 4. Screening laboratory values must be within site normal limits, though trace urine protein is acceptable. -Blood hemoglobin -White blood cell (WBC) count -Neutrophil count -Platelets -Creatinine -AST -ALT -Bilirubin (total) -Glucose (random, must be less than 140) -Urine dipstick for protein and glucose (negative to trace protein are acceptable) -Negative Quantiferon-TB Gold test -Negative HIV 1/2 antibody, (HBsAg), and Hepatitis C virus (HCV) antibody NOTE: See Appendix D for site normal values. Creatinine values lower than the normal range may be acceptable if the PI or a designated licensed clinician determines that these laboratory findings are not clinically significant. HIV and hepatitis C viral load PCR testing may be performed for individuals suspected of having indeterminate antibody testing. For African American participants, a WBC of >/= 3.5 k/mm^3 is acceptable. 5. Able to understand and comply with planned study procedures and willing to be available for all study-required procedures, visits and calls for the duration of the study. 6. Provide written informed consent before initiation of any study procedures. 7. Willing to abstain from donating whole blood or blood derivatives until 90 days after the final study injection.

Exclusion Criteria:

1. History of treatment for active or latent tuberculosis infection or history of positive PPD. 2. History or evidence of active tuberculosis. 3. Has received vaccination or immunotherapy with a BCG product at any time prior to randomization. 4. Shared a residence within the last year prior to randomization with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis. 5. Received a tuberculin skin test within 3 months (90 days) prior to the time of randomization through study day 85. 6. Body temperature >/=100.4°F (>/=38°C) or acute illness within 3 days before study injection days (subject may be rescheduled). 7. A positive serum* or urine pregnancy test at screening or within 24 hours prior to study injection**, women who are planning to become pregnant***, or women who are breastfeeding. * At screening visit only ** If female of childbearing potential as defined in Inclusion Criterion #2 ***from 28 days prior to entering the study until 90 days after the final study injection 8. Immunosuppression as a result of an underlying illness or treatment or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months. 9. An active neoplastic disease* (excluding nonmelanoma skin cancer) or a history of any hematologic malignancy. * defined as neoplastic disease or treatment for neoplastic disease within the past 5 years 10. A history of autoimmune disease (systemic lupus, rheumatoid arthritis, scleroderma, polyarteritis, thyroiditis, etc). 11. Used an immunosuppressive or immunomodulatory drug* for 2 or more consecutive weeks within 6 months prior to the first study injection (nasal and topical steroids are allowed). *such as >0.5 mg/kg/day or >/=20 mg total dose/day of prednisone orally or >800 µg of inhaled beclomethasone 12. A diagnosis of schizophrenia, bipolar disease, or history of hospitalization for a psychiatric condition or previous suicide attempt. 13. A history of treatment for any other psychiatric disorder in the past 3 years that increases the risk to the subject in the opinion of the investigator. 14. A history of receiving immunoglobulin or other blood product within 3 months prior to enrollment through study day 85. 15. Received or plan to receive any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks of any study injection. 16. An acute or chronic medical condition that* would render study injections unsafe or would interfere with the evaluation of responses or is not generally seen in healthy, normal subjects. * in the opinion of the investigator NOTE: This includes, but is not limited to, known cardiac disease, pulmonary disease, liver disease, renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients. 17. History of anaphylaxis or severe allergic reaction to vaccines or history of allergic reaction to eggs, kanamycin-related antibiotics or other components in the antigen and adjuvant formulations. 18. Receipt of an experimental agent* within 1 month before study injections in this study or expectation to receive an experimental agent during the 15-month study period. * vaccine, drug, biologic, device, blood product, or medication 19. Any condition that would* place the subject at an unacceptable injury risk, render him/her unable to meet the requirements of the protocol, or that may interfere with successful study completion. * in the opinion of the investigator 20. A history of alcohol or drug abuse during the previous 1 year* or chronic marijuana abuse or any other illicit drug use. * for example, daily excessive alcohol use or frequ ent binge drinking as determined by the investigator 21. Presence of tattoos that would preclude evaluation of the injection site.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse events considered related to the study injection reported at any point during the study period. | Day 1 through Day 422
The number of subjects experiencing solicited injection site reactions within 7 days following study injection. | 7 days following each study injection
The number of subjects experiencing solicited systemic reactions within 7 days following study injection. | 7 days following each study injection
The number of subjects spontaneously reporting adverse events considered related to the study injection at any point during the study period. | Day 1 through Day 422

SECONDARY OUTCOMES:
Mean fold change from baseline (Day 1) in IgG antibody responses to ID93 on Day 85. | Day 1 and Day 85
Percentage of CD4 and CD8 T cells producing 1 or more cytokines (IFN-gamma, TNF and IL-2) simultaneously in response to stimulation with the ID93 antigen as measured by intracellular cytokine staining at Day 71 relative to baseline (Day 1). | Day 1 and Day 71
The magnitude of Th1 and Th2 cytokine production in PBMCs in response to the ID93 antigen relative to baseline (Day 1) at Day 71, as assayed by Luminex. | Day 1 and Day 71
The proportion of subjects with at least a 4-fold increase in IgG antibody responses to ID93 on Day 85 relative to baseline (Day 1). | Day 1 through Day 85

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa, United States